CLINICAL TRIAL: NCT03558633
Title: A Comparison of the Effects of Cricoid Pressure and Paralaryngeal Pressure to Prevent Regurgitation of Gastric Contents
Brief Title: Cricoid Pressure vs. Paralaryngeal Pressure to Prevent Regurgitation
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, Department of Anesthesiology and Pain medicine, SMG-SNU Boramae Medical Center
Other Study IDs: 20180222/30-2018-11/033
Record Dates: First submitted 2018-04-26; First posted 2018-06-15 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Intubation Complication
Keywords: Cricoid pressure; Paralaryngeal pressure; Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparing the effects of ' Cricoid pressure' or 'Paralaryngeal pressure' during endotracheal intubation procedure.

DETAILED DESCRIPTION:
Applying Cricoid pressure is widely used procedure to prevent gastric contents regurgitation during endotracheal intubation. To find out effectiveness external pressure is applied, the investigators will evaluate the relative position of esophagus and trachea. And also comparing the effects of Cricoid pressure and Paralaryngeal pressure during whole tracheal intubation procedures.

1. Confirm the relative positions between esophagus and trachea in awake patients by using ultrasonography.
2. Compare the effect of 'Cricoid pressure' and 'Paralaryngeal pressure' to esophageal opening during tracheal intubation procedure as below points.

1) Awake states. (Before sedation) 2) Anesthetized states. (After muscle relaxation) 3) During direct intubation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Who would be scheduled any surgery under general anesthesia and agree with the purpose of the study

Exclusion Criteria:

* Diseases or anatomical abnormalities in the neck, larynx, pharynx or esophagus,
* Aspiration tendency
* Known or predicted difficult airway.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Who has any surgery under general anesthesia and agree with the purpose of the study
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Occlusion of esophagus | for 1 minute during direct laryngosopy
  Occlusion of esophagus is checked under the application of cricoid and paralaryngeal pressures during direct laryngsocpy

SECONDARY OUTCOMES:
The relative position of the upper esophageal end to the glottis | 1 minute before and after the induction of anesthesia, during direct laryngoscopy
  The position assessed by using ultrasonography and direct visualization
The outer anteroposterior diameter of the upper esophageal end | During 1 minute in awake and anesthetized paralyzed states
  The outer anteroposterior diameter of the upper esophageal end is assessed before and durng the application of cricoid and paralaryngeal pressures.
POGO score | during direct laryngoscopy
  POGO score under the application of cricoid and paralaryngeal pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Koenig SJ, Lakticova V, Mayo PH. Utility of ultrasonography for detection of gastric fluid during urgent endotracheal intubation. Intensive Care Med. 2011 Apr;37(4):627-31. doi: 10.1007/s00134-010-2125-9. Epub 2011 Feb 2. PMID 21287147